CLINICAL TRIAL: NCT05484466
Title: A Phase IIa Study to Evaluate the Efficacy and Safety of ZM-H1505R in Combination With Entecavir (ETV) Compared With ETV Monotherapy in Patients With Chronic Hepatitis B Who Have Received ETV Monotherapy for at Least 12 Months
Brief Title: A Study to Evaluate the Efficacy and Safety of ZM-H1505R in Combination With ETV Compared With ETV Monotherapy in Patients With CHB
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhimeng Biopharma, Inc. (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZM-H1505R-201
Record Dates: First submitted 2022-07-20; First posted 2022-08-02 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2022-07

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B, Chronic; Multicenter; Randomized; Double-Blind; Placebo-Controlled; Phase IIa
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Intervention Model Description: The study is planned to enroll 90 adult CHB subjects who have received ETV monotherapy for at least 12 months and are still receiving ETV monotherapy (0.5 mg, QD) continuously. Eligible subjects will be randomized in a 1:1:1 ratio into 3 treatment groups. Both HBeAg positive and negative subjects will be included. There will be 20 HBeAg positive subjects and 10 HBeAg negative subjects in each treatment group. The treatment regimens in each group are as follows:
  Group A: ZM-H1505R 50 mg QD + Baraclude 0.5 mg QD Group B: ZM-H1505R 100 mg QD + Baraclude 0.5 mg QD Group C: ZM-H1505R placebo QD + Baraclude 0.5 mg QD After 48 weeks of treatment with the corresponding regimen, subjects will continue to take Baraclude 0.5 mg QD, as a monotherapy for a 12-week follow-up period for observation of efficacy and safety of ZM-H1505R.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A:ZM-H1505R 50 mg QD + Baraclude 0.5 mg QD (Experimental): The treatment regimen is as follow:
  Group A: ZM-H1505R 50 mg QD + Baraclude 0.5 mg QD 48weeks After 48 weeks of treatment with the corresponding regimen, subjects will continue to take Baraclude 0.5 mg QD, as a monotherapy for a 12-week .
  Interventions: Drug: ZM-H1505R; Other: ZM-H1505R placebo; Combination Product: Baraclude
- Group B:ZM-H1505R 100 mg QD + Baraclude 0.5 mg QD (Experimental): The treatment regimen is as follow:
  Group B: ZM-H1505R 100 mg QD + Baraclude 0.5 mg QD 48weeks After 48 weeks of treatment with the corresponding regimen, subjects will continue to take Baraclude 0.5 mg QD, as a monotherapy for a 12-week .
  Interventions: Drug: ZM-H1505R; Combination Product: Baraclude
- Group C:ZM-H1505R placebo QD + Baraclude 0.5 mg QD (Placebo Comparator): The treatment regimen is as follow:
  Group C: ZM-H1505R placebo QD + Baraclude 0.5 mg QD 48weeks After 48 weeks of treatment with the corresponding regimen, subjects will continue to take Baraclude 0.5 mg QD, as a monotherapy for a 12-week .
  Interventions: Other: ZM-H1505R placebo; Combination Product: Baraclude

INTERVENTIONS:
Drug: ZM-H1505R — There are three groups in this study. ZM-H1505R will be used in group A and Group B ，Subjects can use it for 48 weeks Group A: 30 subjects； ZM-H1505R 50 mg QD +ZM-H1505R placebo； Group B: 30 subjects； ZM-H1505R 100 mg QD
  Arms: Group A:ZM-H1505R 50 mg QD + Baraclude 0.5 mg QD; Group B:ZM-H1505R 100 mg QD + Baraclude 0.5 mg QD
Other: ZM-H1505R placebo — There are three groups in this study. ZM-H1505R will be used in group A and Group C ，Subjects can use it for 48 weeks Group A: 30 subjects；ZM-H1505R 50 mg +ZM-H1505R placebo 50mg QD ； Group C: 30 subjects；ZM-H1505R placebo 100mg QD
  Arms: Group A:ZM-H1505R 50 mg QD + Baraclude 0.5 mg QD; Group C:ZM-H1505R placebo QD + Baraclude 0.5 mg QD
Combination Product: Baraclude — All subjects were orally administered once a day at night ： Baraclude® 0.5 mg QD，60weeks

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled phase IIa study, designed to evaluate the efficacy and safety of ZM-H1505R in combination with Baraclude versus Baraclude monotherapy in adult CHB subjects with HBV DNA <2000 IU/mL but ≥ 50 IU/mL and who have received ETV (0.5 mg, once daily [QD)] monotherapy for at least 12 months.

The study is planned to enroll 90 adult CHB subjects who have received ETV monotherapy for at least 12 months and are still receiving ETV monotherapy (0.5 mg, QD) continuously. Eligible subjects will be randomized in a 1:1:1 ratio into 3 treatment groups. Both HBeAg positive and negative subjects will be included. There will be 20 HBeAg positive subjects and 10 HBeAg negative subjects in each treatment group.

After 48 weeks of treatment with the corresponding regimen, subjects will continue to take Baraclude 0.5 mg QD, as a monotherapy for a 12-week follow-up period for observation of efficacy and safety of ZM-H1505R.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled phase IIa study, designed to evaluate the efficacy and safety of ZM-H1505R in combination with Baraclude versus Baraclude monotherapy in adult CHB subjects with HBV DNA <2000 IU/mL but ≥ 50 IU/mL and who have received ETV (0.5 mg, once daily [QD)] monotherapy for at least 12 months.

The study is planned to enroll 90 adult CHB subjects who have received ETV monotherapy for at least 12 months and are still receiving ETV monotherapy (0.5 mg, QD) continuously. Eligible subjects will be randomized in a 1:1:1 ratio into 3 treatment groups. Both HBeAg positive and negative subjects will be included. There will be 20 HBeAg positive subjects and 10 HBeAg negative subjects in each treatment group. The treatment regimens in each group are as follows:

Group A: ZM-H1505R 50 mg QD + Baraclude 0.5 mg QD Group B: ZM-H1505R 100 mg QD + Baraclude 0.5 mg QD Group C: ZM-H1505R placebo QD + Baraclude 0.5 mg QD After 48 weeks of treatment with the corresponding regimen, subjects will continue to take Baraclude 0.5 mg QD, as a monotherapy for a 12-week follow-up period for observation of efficacy and safety of ZM-H1505R.

ELIGIBILITY:
Inclusion criteria

* 1.Able to understand and sign the written informed consent form (the informed consent should be obtained prior to any study procedure);
* 2.Males and females aged 18-65 (inclusive);
* 3.Have been used ETV (0.5 mg, QD) monotherapy for at least 12 months at the time of screening; and able to provide evidence of existing HBV infection (e.g., HBsAg and/or HBV DNA positive), or HBsAg positive at screening;
* 4.Plasma HBV DNA < 2000 IU/mL but ≥ 50 IU/mL in 2 consecutive tests at least 30 days apart during the screening period (serum samples will be delivered to the designated central laboratory for testing)
* 5.Women of childbearing potential or males with female partners of childbearing potential must agree to voluntarily use the contraceptive methods specified in the protocol from screening to 28 days after the last dose of the study (see Appendix 1).

Exclusion criteria

* 1.Progressive fibrosis or cirrhosis detected at screening, or progressive fibrosis or cirrhosis defined as follows: Metavir ≥ 3 or Ishak fibrosis score ≥ 4 by liver biopsy within 1 year prior to screening; or in the absence of an appropriate liver biopsy, liver stiffness test (FibroScan)

  ≥ 9 kPa within 3 months prior to screening;
* 2.History of hepatocellular carcinoma (HCC); or serum alpha-fetoprotein (AFP) ≥ 50 ng/mL at screening, or imaging examination such as abdominal ultrasound, CT (computed tomography) or MRI (magnetic resonance imaging) suggesting possible HCC;
* 3.Subjects meeting any of the following clinical laboratory parameters at screening:

  1. Hemoglobin < 120 g/L (for males) or < 110 g/L (for females);
  2. Platelet count < 100 × 109/L;
  3. Neutrophil count < 1.5 × 109/L;
  4. Alanine aminotransferase (ALT) > 3 × upper limit of normal (×ULN);
  5. International normalized ratio (INR) of prothrombin time > 1.3;
  6. Albumin < 35 g/L;
  7. Total bilirubin > 2 × ULN, and direct bilirubin > 1.5 × ULN;
  8. Estimated glomerular filtration rate < 60 mL/min/1.73 m2 (calculated using the CKD-MDRD formula, see Appendix 2).
* 4.Abnormal result of electrocardiogram (ECG) at screening and inappropriate for the study participation judged by the investigator; Or QTcF (QT corrected using the Fridericia formula): > 450 ms for males, > 470 ms for females at screening;
* 5.Co-infection with human immunodeficiency virus (HIV), hepatitis A virus (HAV), hepatitis C virus (HCV), hepatitis D virus (HDV) or hepatitis E virus (HEV); Note: Subjects with positive HCV antibody (Ab) but negative HCV RNA and subjects with positive HEV immunoglobulin M (IgM) but negative HEV RNA will NOT be excluded.
* 6.Other malignancy unless the subject's malignancy has been cured by surgical resection (e.g., basal cell skin cancer); Note: Subjects who are suspected of having malignancy must be excluded regardless of evidence of local recurrence or metastasis.
* 7.History of chronic liver disease with a non-HBV etiology, such as alcoholic liver disease, autoimmune liver disease, hereditary liver disease, non-alcoholic fatty liver disease, except for simple fatty liver disease;
* 8.Other concurrent severe systemic diseases or clinical manifestations, for which the investigator considers not suitable to participate in this study, including but not limited to:

  1. Circulatory system diseases: such as unstable angina, myocardial infarction, congestive heart failure, and poorly controlled or refractory hypertension (for example, after medication treatment, systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg);
  2. Respiratory system diseases: such as severe chronic obstructive pulmonary disease;
  3. Primary or secondary renal diseases (such as chronic renal decompensation and renal diseases associated with diabetes, hypertension, and vascular diseases);
  4. Endocrine system diseases: such as poorly controlled diabetes or thyroid disease;
  5. Autoimmune diseases: such as systemic lupus erythematosus, idiopathic thrombocytopenic purpura, rheumatoid arthritis, inflammatory bowel disease, sarcoidosis, autoimmune hemolytic anemia, and psoriasis;
  6. Neuropsychiatric diseases: such as epilepsy, schizophrenia, and depression;
* 9.Use of any investigational product or drug not approved by regulatory authorities within 3 months prior to screening;
* 10.History of persistent alcohol comsumption (alcohol consumption exceeding 40 g ethanol for males or 20 g ethanol for females per day on average) within 6 months prior to screening;
* 11.History of drug dependence or drug abuse;
* 12.Pregnant or breastfeeding women;
* 13.Known hypersensitivity to the active ingredient or formulation excipients of the investigational drug;
* 14.Inappropriate for the study participation for any reason not otherwise listed as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects who achieves complete virologic response (CVR) at week 24 of treatment period. | 24 weeks
  To evaluate the efficacy of ZM-H1505R in combination with ETV (Baraclude®) versus Baraclude® monotherapy in adult CHB subjects who have received ETV monotherapy for at least 12 months.
  Percentage of subjects who achieves complete virologic response (CVR) at week 24 of treatment period.
  (CVR is defined as HBV DNA ≤ 10 IU/mL.)
To evaluate the safety of ZM-H1505R in combination with Baraclude versus Baraclude monotherapy in adult CHB subjects who have received ETV monotherapy for at least 12 months. | 24 weeks
  An AE was any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE was any unfavorable and unintended sign, symptom, disease, and/or laboratory or physiological observation that may or may not be related to the investigational medicinal product.

SECONDARY OUTCOMES:
To evaluate the long-term safety of ZM-H1505R in combination with Baraclude® versus Baraclude® monotherapy in adult CHB subjects who have received ETV monotherapy for at least 12 months. | 60 weeks
  An AE was any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE was any unfavorable and unintended sign, symptom, disease, and/or laboratory or physiological observation that may or may not be related to the investigational medicinal product.
Percentage of subjects who achieves CVR at each scheduled visits other than week 24 visit | 60 weeks
  To evaluate the long-term safety of ZM-H1505R in combination with Baraclude versus Baraclude® monotherapy in adult CHB subjects who have received ETV monotherapy for at least 12 months.
  Percentage of subjects who achieves CVR at each scheduled visits other than week 24 visit.
  (CVR is defined as HBV DNA ≤ 10 IU/mL.)
Time to achieve CVR in each group | 60 weeks
  To evaluate other virology indicators of ZM-H1505R in combination with Baraclude versus Baraclude monotherapy in adult CHB subjects who have received ETV monotherapy for at least 12 months.
  Time to achieve CVR in each group (CVR is defined as HBV DNA ≤ 10 IU/mL.)
Changes from baseline in quantitative HBV ribonucleic acid (RNA) at each scheduled visits | Baseline, Week 24, Week 48 and Week 60
  Change in Mean log10 HBV RNA From Baseline (Day -60 to Day -1) to Week 24, Week 48, or Week 60 on ZM-H1505R + SOC ETV as Compared to Placebo + SOC ETV Hepatitis B virus (HBV) RNA was measured using COBAS 6800. The lower limit of quantitation (LLOQ) was 10 Copies/mL.
Percentage of subjects whose quantitative HBV RNA is ≤ 10 copies/mL at each scheduled visits | 60 weeks
  To evaluate other virology indicators of ZM-H1505R in combination with Baraclude versus Baraclude monotherapy in adult CHB subjects who have received ETV monotherapy for at least 12 months.
  Percentage of subjects whose quantitative HBV RNA is ≤ 10 copies/mL at each scheduled visits
Changes from baseline in quantitative hepatitis B surface antigen (HBsAg) at weeks 4, 12, 24, 36, 48, and 60 | Baseline;at weeks 4, 12, 24, 36, 48, and 60
  To evaluate other virology indicators of ZM-H1505R in combination with Baraclude versus Baraclude monotherapy in adult CHB subjects who have received ETV monotherapy for at least 12 months.
  Changes from baseline in quantitative hepatitis B surface antigen (HBsAg) at weeks 4, 12, 24, 36, 48, and 60
Percentage of subjects achieving HBsAg loss at weeks 24, 48, and 60 | At weeks 24, 48, and 60
  To evaluate other virology indicators of ZM-H1505R in combination with Baraclude versus Baraclude monotherapy in adult CHB subjects who have received ETV monotherapy for at least 12 months.
  6) Percentage of subjects achieving HBsAg loss at weeks 24, 48, and 60; (HBsAg loss is defined as HBsAg positive before treatment and HBsAg negative after treatment.)
Percentage of subjects achieving HBsAg seroconversion at weeks 24, 48, and 60 | At weeks 24, 48, and 60
  To evaluate other virology indicators of ZM-H1505R in combination with Baraclude versus Baraclude monotherapy in adult CHB subjects who have received ETV monotherapy for at least 12 months.
  Percentage of subjects achieving HBsAg seroconversion at weeks 24, 48, and 60; (HBsAg seroconversion is defined as HBsAg positive before treatment and HBsAg negative after treatment, with hepatitis B surface antibody [HBsAb] changed to positive.)
Percentage of subjects achieving hepatitis B e antigen (HBeAg) loss at weeks 24, 48, and 60 | At weeks 24, 48, and 60
  To evaluate other virology indicators of ZM-H1505R in combination with Baraclude versus Baraclude monotherapy in adult CHB subjects who have received ETV monotherapy for at least 12 months.
  Percentage of subjects achieving hepatitis B e antigen (HBeAg) loss at weeks 24, 48, and 60 (only for subjects who are HBeAg positive at baseline); (HBeAg loss is defined as a subject who is HBeAg positive before treatment and becomes HBeAg negative after treatment.)
Percentage of subjects with HBeAg seroconversion at weeks 24, 48, and 60 | At weeks 24, 48, and 60
  To evaluate other virology indicators of ZM-H1505R in combination with Baraclude versus Baraclude monotherapy in adult CHB subjects who have received ETV monotherapy for at least 12 months.
  Percentage of subjects with HBeAg seroconversion at weeks 24, 48, and 60 (only for subjects who are HBeAg positive at baseline); (HBeAg seroconversion is defined as HBeAg positive before treatment and HBeAg negative after treatment, with hepatitis B e antibody [HBeAb] changed to positive.)
Changes from baseline in quantitative hepatitis B core-related antigen (HBcrAg) at weeks 4, 12, 24, 36, 48, and 60 | Baseline；at weeks 4, 12, 24, 36, 48, and 60
  To evaluate other virology indicators of ZM-H1505R in combination with Baraclude versus Baraclude monotherapy in adult CHB subjects who have received ETV monotherapy for at least 12 months.
  Changes from baseline in quantitative hepatitis B core-related antigen (HBcrAg) at weeks 4, 12, 24, 36, 48, and 60
THBV genotypic resistance. | 60 weeks
  The number of cases and percentages of subjects with HBV genotypic resistance.
Plasma concentration of ZM-H1505R | Baseline；at weeks 4, 12, 24, 36, 48
  For determination of ZM-H1505R plasma concentration, sparse PK blood samples will be collected in all subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No